CLINICAL TRIAL: NCT06798987
Title: Characterization of the Spatial Distribution and Drivers of the Association of Meteorological Factors and Air Pollution with the Number of First Aiders
Brief Title: Based on the Data from the Zhejiang Emergency Center, Explore the Independent and Interactive Effects of the Association Between Meteorological Factors and Air Pollution and the Number of Emergency Personnel, Identify the Relevant Vulnerable Population Characteristics, Sensitive Disease Types
Status: Enrolling by invitation | Type: Observational
Sponsor: Li hengjie (Other)
Responsible Party: Sponsor-Investigator, Li hengjie, Protomedicus, Zhejiang Provincial People's Hospital
Organization: Zhejiang Provincial People's Hospital (Other)
Other Study IDs: QT202146
Record Dates: First submitted 2025-01-13; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Fig. Impetuous
MeSH Terms: interventions — Air Pollution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: Meteorological conditions and air pollution — Climate change e.g. global surface temperature rise; extreme weather events e.g. heat waves, floods

SUMMARY:
Based on the health data from Zhejiang Emergency Command Center, combined with meteorological, air pollution, land use and socio-economic data of Zhejiang Province, distributional lag nonlinear models, grouped weighted quantile and regression and Bayesian spatial models were used to explore the independent and interactive effects of the association between meteorological factors and air pollution and the number of first-aiders, to identify the related characteristics of the vulnerable populations, the types of sensitive diseases and the high-risk areas, and to elucidate the driving factors of the association between meteorological factors and air pollution and the number of first-aiders. It also clarifies the drivers of the association between meteorological factors and air pollution and the number of emergencies, so as to provide a reference for the government to take targeted measures to reduce the burden of related healthcare services.

ELIGIBILITY:
Inclusion Criteria:

-Emergency data of Zhejiang Emergency Command Center in the past 5 years

Exclusion Criteria:

* Prehospital emergency information from non-Zhejiang province domains
* Emergency calls due to labor and delivery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Number of emergency patients per hour at the emergency command center of Zhejiang Province
Sampling Method: Non-Probability Sample
Enrollment: 1500000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of first aiders per hour as assessed by R4.4.0 | 6 months
Vulnerable population characteristics as assessed by R4.4.0 | 6 Months
Types of Sensitive Diseases as assessed by R4.4.0 | 6 Month
High-risk areas as assessed by R4.4.0 | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, China

REFERENCES:
- [Background] Cui Y, Ai S, Liu Y, Qian ZM, Wang C, Sun J, Sun X, Zhang S, Syberg KM, Howard S, Qin L, Lin H. Hourly associations between ambient temperature and emergency ambulance calls in one central Chinese city: Call for an immediate emergency plan. Sci Total Environ. 2020 Apr 1;711:135046. doi: 10.1016/j.scitotenv.2019.135046. Epub 2019 Nov 3. PMID 31812379
- [Background] Bobb JF, Peng RD, Bell ML, Dominici F. Heat-related mortality and adaptation to heat in the United States. Environ Health Perspect. 2014 Aug;122(8):811-6. doi: 10.1289/ehp.1307392. Epub 2014 Apr 29. PMID 24780880
- [Background] Phosri A, Ueda K, Seposo X, Honda A, Takano H. Effect modification by temperature on the association between O3 and emergency ambulance dispatches in Japan: A multi-city study. Sci Total Environ. 2023 Feb 25;861:160725. doi: 10.1016/j.scitotenv.2022.160725. Epub 2022 Dec 6. PMID 36493818
- [Background] Wang X, Leng M, Liu Y, Qian ZM, Zhang J, Li Z, Sun L, Qin L, Wang C, Howard SW, Vaughn MG, Yan Y, Lin H. Different sized particles associated with all-cause and cause-specific emergency ambulance calls: A multicity time-series analysis in China. Sci Total Environ. 2021 Aug 20;783:147060. doi: 10.1016/j.scitotenv.2021.147060. Epub 2021 Apr 18. PMID 34088160
- [Background] Michikawa T, Sasaki J, Yamazaki S, Takami A, Asakura K, Imamura H, Ueda K, Saito S, Hoshi J, Yoshino A, Sugata S, Nitta H, Nishiwaki Y. A Case-Crossover Analysis of the Association between Exposure to Total PM2.5 and Its Chemical Components and Emergency Ambulance Dispatches in Tokyo. Environ Sci Technol. 2022 Jun 7;56(11):7319-7327. doi: 10.1021/acs.est.1c08219. Epub 2022 May 24. PMID 35608996
- [Background] Dawson LP, Andrew E, Nehme Z, Bloom J, Cox S, Anderson D, Stephenson M, Lefkovits J, Taylor AJ, Kaye D, Guo Y, Smith K, Stub D. Temperature-related chest pain presentations and future projections with climate change. Sci Total Environ. 2022 Nov 20;848:157716. doi: 10.1016/j.scitotenv.2022.157716. Epub 2022 Jul 29. PMID 35914598
- [Background] Sangkharat K, Mahmood MA, Thornes JE, Fisher PA, Pope FD. Impact of extreme temperatures on ambulance dispatches in London, UK. Environ Res. 2020 Mar;182:109100. doi: 10.1016/j.envres.2019.109100. Epub 2020 Jan 3. PMID 31918315
- [Background] Chen R, Yin P, Wang L, Liu C, Niu Y, Wang W, Jiang Y, Liu Y, Liu J, Qi J, You J, Kan H, Zhou M. Association between ambient temperature and mortality risk and burden: time series study in 272 main Chinese cities. BMJ. 2018 Oct 31;363:k4306. doi: 10.1136/bmj.k4306. PMID 30381293
- [Background] Gasparrini A, Guo Y, Hashizume M, Lavigne E, Zanobetti A, Schwartz J, Tobias A, Tong S, Rocklov J, Forsberg B, Leone M, De Sario M, Bell ML, Guo YL, Wu CF, Kan H, Yi SM, de Sousa Zanotti Stagliorio Coelho M, Saldiva PH, Honda Y, Kim H, Armstrong B. Mortality risk attributable to high and low ambient temperature: a multicountry observational study. Lancet. 2015 Jul 25;386(9991):369-75. doi: 10.1016/S0140-6736(14)62114-0. Epub 2015 May 20. PMID 26003380
- [Background] Ahn J, Bae S, Chung BH, Myong JP, Park MY, Lim YH, Kang MY. Association of summer temperatures and acute kidney injury in South Korea: a case-crossover study. Int J Epidemiol. 2023 Jun 6;52(3):774-782. doi: 10.1093/ije/dyac163. PMID 35950799
- [Background] Achilleos S, Al-Ozairi E, Alahmad B, Garshick E, Neophytou AM, Bouhamra W, Yassin MF, Koutrakis P. Acute effects of air pollution on mortality: A 17-year analysis in Kuwait. Environ Int. 2019 May;126:476-483. doi: 10.1016/j.envint.2019.01.072. Epub 2019 Mar 4. PMID 30844583
- [Background] Fiore AM, Naik V, Spracklen DV, Steiner A, Unger N, Prather M, Bergmann D, Cameron-Smith PJ, Cionni I, Collins WJ, Dalsoren S, Eyring V, Folberth GA, Ginoux P, Horowitz LW, Josse B, Lamarque JF, MacKenzie IA, Nagashima T, O'Connor FM, Righi M, Rumbold ST, Shindell DT, Skeie RB, Sudo K, Szopa S, Takemura T, Zeng G. Global air quality and climate. Chem Soc Rev. 2012 Oct 7;41(19):6663-83. doi: 10.1039/c2cs35095e. Epub 2012 Aug 6. PMID 22868337
- [Background] Chen K, Wolf K, Breitner S, Gasparrini A, Stafoggia M, Samoli E, Andersen ZJ, Bero-Bedada G, Bellander T, Hennig F, Jacquemin B, Pekkanen J, Hampel R, Cyrys J, Peters A, Schneider A; UF&HEALTH Study Group. Two-way effect modifications of air pollution and air temperature on total natural and cardiovascular mortality in eight European urban areas. Environ Int. 2018 Jul;116:186-196. doi: 10.1016/j.envint.2018.04.021. Epub 2018 Apr 22. PMID 29689465
- [Background] Doherty RM, Heal MR, O'Connor FM. Climate change impacts on human health over Europe through its effect on air quality. Environ Health. 2017 Dec 5;16(Suppl 1):118. doi: 10.1186/s12940-017-0325-2. PMID 29219103
- [Background] Ebi KL, Capon A, Berry P, Broderick C, de Dear R, Havenith G, Honda Y, Kovats RS, Ma W, Malik A, Morris NB, Nybo L, Seneviratne SI, Vanos J, Jay O. Hot weather and heat extremes: health risks. Lancet. 2021 Aug 21;398(10301):698-708. doi: 10.1016/S0140-6736(21)01208-3. PMID 34419205
- [Background] Khoshakhlagh AH, Mohammadzadeh M, Gruszecka-Kosowska A, Oikonomou E. Burden of cardiovascular disease attributed to air pollution: a systematic review. Global Health. 2024 May 3;20(1):37. doi: 10.1186/s12992-024-01040-0. PMID 38702798